CLINICAL TRIAL: NCT05212649
Title: Optimizing Risk Stratification in Predicting Poor Prognosis in Post-Acute Heart Failure With Reduced Ejection Fraction
Brief Title: Optimized Peak VO2 in Predicting Advanced HF
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202001285B0D001
Record Dates: First submitted 2022-01-03; First posted 2022-01-28 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure; Morality; Transplant; Failure, Heart
Keywords: advance heart failure; cardiac transplantation; Peak oxygen consumption; Guideline-directed medical therapy; Risk score; Heart Failure Survival Score
MeSH Terms: conditions — Heart Failure | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- More-GDMT: Baseline guideline-directed medications therapy (GDMT), including angiotensin-converting enzyme inhibitors (ACEI) or angiotensin II receptor blocker (ARB), beta-blockers, mineralocorticoid receptor antagonist (MRA), and angiotensin receptor neprilysin inhibitor (ARNI) were documented at discharge. More-GDMT group was defined as patient population received GDMT >=2 kinds of above medications.
  Interventions: Diagnostic Test: cardiopulmonary exercise test
- Few-GDMT group: Baseline guideline-directed medications therapy (GDMT), including angiotensin-converting enzyme inhibitors (ACEI) or angiotensin II receptor blocker (ARB), beta-blockers, mineralocorticoid receptor antagonist (MRA), and angiotensin receptor neprilysin inhibitor (ARNI) were documented at discharge. Few GDMT-group was defined as patients who received GDMT < 2 kinds of the above medications.
  Interventions: Diagnostic Test: cardiopulmonary exercise test

INTERVENTIONS:
Diagnostic Test: cardiopulmonary exercise test — CPET was performed in this HF cohort within one month after being discharged and interpreted as previously described. Patients underwent an upright graded cycle ergometer exercise using a personalized ramp protocol or a motorized treadmill using a modified Bruce or Cornell protocol. Peak VO2 data measured by cycle ergometer were increased by 10% to allow a comparison between the two different procedures. Peak VO2 was defined as the highest 30-second average value obtained during exercise. Submaximal CPET variables such as ventilatory efficiency were calculated by the slope of VE versus VCO2 below the ventilatory compensatory point (VCP). If the slope of VE/VCO2 can't be calculated, we used the nadir of VE/VCO2, or the ratio of VE/VCO2 at the anaerobic threshold (AT) as the variable of ventilatory efficiency. The AT was determined by the V-slope method.

SUMMARY:
The ability and timely selection of severe heart failure (HF) patients for cardiac transplantation and advanced HF therapy is challenging. Peak VO2 by cardiopulmonary exercise test (CPET) was used for transplant listing. This study aimed to reassess the prognostic significance of peak VO2 and to compare that with the Heart Failure Survival Score in the current optimized novel guideline-directed medical therapy (GDMT).

DETAILED DESCRIPTION:
Investigators retrospectively collected acute HF patients discharged alive from the hospital. Investigators divided participants into more-GDMT (≥2 kinds) and few-GDMT (<2 kinds) groups and compared the prognostic significance of peak VO2 and HFSS for combined all-cause mortality and urgent cardiac transplantation.

ELIGIBILITY:
Inclusion Criteria:

* acute HF patients with reduced ejection fraction (left ventricular ejection fraction, LVEF <=40%) and discharged alive from the hospital
* patients with age >= 20 years of age
* patients who performed cardiopulmonary exercise test (CPET) within one month after discharge
* patients with serum B-type natriuretic peptide (BNP) level >100 pg/mL.

Exclusion Criteria:

* patients with estimated survival time < 6 months
* patients who could not tolerate exercise test due to muscular-skeletal disorder or other reason
* patients who had severe valvular heart disease.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators retrospectively collected acute HF patients discharged alive from the hospital. Investigators divided participants into more-GDMT (>= 2 kinds) and few-GDMT (<2 kinds) groups and compared the prognostic significance of peak VO2 and Heart Failure Survival Score for combined all-cause mortality and urgent cardiac transplantation.
Sampling Method: Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | May, 2014 ~ June 2020
  Number of participants that had occurrence of the mortality which is defined as all-cause mortality
urgent heart transplant | May, 2014 ~ June 2020
  Number of participants that had occurrence of the urgent heart transplant

CONTACTS AND LOCATIONS:
Overall Officials: Shyh-Ming Chen, MD, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang Gung Memorial Hospital Heart Failure Center, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data sharing plans will be discussed with other investigators